CLINICAL TRIAL: NCT01080950
Title: Vitamin d and Zinc Levels in Patients With Fever
Brief Title: Vitamin D Zinc Fever
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: renana shor md, Assaf - Harofeh MC
Other Study IDs: vitamin d zinc and fever
Record Dates: First submitted 2010-03-03; First posted 2010-03-05 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2010-03

CONDITIONS: Sepsis; Fever; Vitamin D
Keywords: zinc; sepsis; fever; vitamin d
MeSH Terms: conditions — Sepsis; Fever

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood drawn for vitamin d will be freezed and stored until all samples have been collected and only than will it be analyzed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- fever zinc vit. d: patients with fever but without sepsis
- sepsis zinc vit. d: patients with sepsis

SUMMARY:
Zinc and vitamin d deficiency are associated with a state of inflammation/atherosclerosis.

There are studies demonstrating an association between vitamin d deficiency and respiratory illnesses.

Both zinc and vitamin d are associated with oxidative stress and inflammation.

DETAILED DESCRIPTION:
Both vit. d and zinc share anti inflammatory and anti oxidative actions. vit. d deficiency is associated with an increase in serum levels of proinflammatory cytokines and decreased levels of anti inflammatory cytokines.

there are reports concerning the association of vit. d deficiency with infections.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years

Exclusion Criteria:

* CCT<90
* taking calcium
* hyper/hypoparathyroidism
* active malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients hospitalized with fever and or sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofeh Mc, Ẕerifin, Israel